CLINICAL TRIAL: NCT00142493
Title: Effect of Affective Content on Drug Induced Amnesia of Episodic Memory
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-087
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Memory Losses; Amnesia-Memory Loss
Keywords: Episodic Memory; Amnesia; Amnesia, Temporary
MeSH Terms: conditions — Memory Disorders; Amnesia | interventions — Propofol; Thiopental; Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Propofol
- 2 (Experimental)
  Interventions: Drug: Thiopental Sodium
- 3 (Experimental)
  Interventions: Drug: Dexmedetomidine Hydrochloride
- 4 (Experimental)
  Interventions: Drug: Midazolam Hydrochloride
- 5 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Propofol — 1.2ug/ml
  Arms: 1
Drug: Thiopental Sodium — 2.0ug/ml
  Arms: 2
Drug: Dexmedetomidine Hydrochloride — 0.5ng/ml
  Arms: 3
Drug: Midazolam Hydrochloride — 60ng/ml
  Arms: 4
Drug: placebo — intralipid, saline, saline with multi-Vit solution
  Arms: 5

SUMMARY:
The purpose of this research is to understand how some of the drugs commonly used in anesthesia impair memory. We are particularly interested in whether the emotion associated with a memory influences how well these drugs are able to block memory. We are studying four commonly used drugs-propofol, thiopental, midazolam, and dexmedetomidine, all of which may have slightly differing effects. We will also study an inactive substance, called a placebo, that should have no effect. The results of this study will provide information that will be useful in understanding how memory works, how these drugs affect memory, and possibly why some people don't have their memory blocked as easily as others.

DETAILED DESCRIPTION:
The protocol "Effect of Affective Content on Drug Induced Amnesia of Episodic Memory" investigates the relationship between the ability of affective ('emotional') content to modulate the formation of episodic memory, and the memory impairment ('amnestic') effects of several common intravenous anesthetic drugs. Because memory modulation by affective content appears to be a distinct memory process, the underlying question is whether drugs that impair memory via different mechanisms will have differing effects on memory modulation. Specifically, the objectives are: (1) To study the influence of three GABAergic agents (thiopental, propofol, and midazolam) and one α2-adrenergic agent (dexmedetomidine) on the ability of affective content to modulate the strength of episodic memory; and (2) To study whether the subliminal ('consciously imperceptible') presentation of emotional words can influence memory for visual stimuli shown immediately after the subliminal presentation.

A maximum of eighty volunteers will receive sub-anesthetic doses of one of the four study drugs, or placebo, while performing a visual continuous recognition task ('CRT') of pictures with randomly varying affective load. Drug effect on affective modulation of working and early long-term memory behavior will be examined by analyzing which images are and are not recognized during the CRT. Drug effect on affective modulation of later long-term memory will be examined by analyzing which images are recognized several hours after presentation.

In a second experiment, emotive and non-emotive words are subliminally presented immediately before the presentation of a 'bland' picture. The ability of the subliminally presented word to influence memory will be examined by analyzing which bland images are recognized several hours later.

Three hypotheses are tested:

The memory impairment effected by GABAergic drugs will be stronger for memory of emotively positive images than for memory of emotively negative images

The memory impairment effected by dexmedetomidine will be similar for memory of emotively positive and negative images

Recognition memory for neutral, non-arousing images will be greater if the image is immediately preceded by the subliminal presentation of an emotively arousing word than if it is preceded by an emotively non-arousing word

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal volunteers, age 18 to 50 years *,who show no evidence of neurologic deficit on questionnaire and physical examination.
* Females must be non-pregnant as demonstrated using a serum pregnancy test.
* Right hand dominant.
* High school education or above.
* English as native language or equivalent degree of fluency. *Age group selected based on pharmacokinetic models for drug infusion, and norms for standardized memory tests.

Exclusion Criteria:

* Any evidence of neurologic deficit including seizures, severe head trauma resulting in unconsciousness, or any previously abnormal study of CNS - (e.g. MRI, EEG, etc.)
* Any deficit in auditory or visual ability.
* Any history of hypertension (resting BP >150 systolic, >100 diastolic) or taking anti- hypertensive medication or cardiovascular disease.
* Significant pulmonary, renal, gastrointestinal, or endocrine metabolic disease which in the opinion of the investigator would complicate the goals of this study.
* Allergy to propofol or eggs.
* History of acute intermittent porphyria in subject or subject's blood relatives.
* History of substance abuse
* Currently taking centrally acting medications (e,g, benzodiazepines or anti depressants)
* Subjects whose body weight relative to their height exceeds accepted criteria for defining obesity in the general population (Body Mass Index > 30). Excess weight can affect the pharmacodynamics of the drug in the body.
* Anyone who, in the opinion of the investigators, would be unwilling or unable to tolerate the procedures and/or comply with the task instructions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2004-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To study the influence of three GABAergic agents (thiopental, propofol, and midazolam) and one α2-adrenergic agent (dexmedetomidine) on the ability of affective content to modulate the strength of episodic memory | over a two day period

SECONDARY OUTCOMES:
To study whether the subliminal ('consciously imperceptible') presentation of emotional words can influence memory for visual stimuli shown immediately after the subliminal presentation | over a two day period

CONTACTS AND LOCATIONS:
Overall Officials: Kane O. Pryor, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org